CLINICAL TRIAL: NCT06765603
Title: Evaluating the Efficacy of the Combination of Multi-zonal Contact Lens and Atropine for Controlling Myopia Progression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Audrey Wei-Lin Chia, pi, Singapore National Eye Centre
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1867/109/2021
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: myopia intervention
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Atropine - SVCL (Experimental): Atropine 0.025%
  Interventions: Drug: Atropine 0.025%; Device: Single vision Contact lens
- Atropine- multizonal CL (Active Comparator): Atropine 0.025% and multizonal CL
  Interventions: Drug: Atropine 0.025%; Device: Multizonal contact lens
- Multizonal CL - placebo drop (Active Comparator): Multizonal CL
  Interventions: Device: Multizonal contact lens; Drug: Placebo
- Placebo drop and SVCL (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Device: Single vision Contact lens

INTERVENTIONS:
Drug: Atropine 0.025% — Atropine 0.025%
  Arms: Atropine - SVCL; Atropine- multizonal CL
Device: Multizonal contact lens — Multizonal CL
  Arms: Atropine- multizonal CL; Multizonal CL - placebo drop
Drug: Placebo — Placebo
  Arms: Multizonal CL - placebo drop; Placebo drop and SVCL
Device: Single vision Contact lens — Single vision contact lens
  Arms: Atropine - SVCL; Placebo drop and SVCL

SUMMARY:
The aim of the study is to explore efficacy of combination Atropine and multifocal CL. Randomized Control Trial including 4 arms: Atropine / multizonal CL; Atropine/ SV CL, Placebo drop/ multizonal CL; Placebo drop/ SV CL. Followed over 1 year with outcome measure of change in spherical equivalent and axial length.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Between 7 and 12 (inclusive) years of age at the time of screening.
* spherical equivalent of cycloplegic objective refraction (by autorefraction) range of -0.75 D to -4.50 D (inclusive) in each eye.
* Refractive cylinder less than 1.12 D (inclusive)
* Best-corrected visual acuity (BCVA) of 0.04 logMAR or better in each eye, with difference less than 0.20 logMAR between eyes.
* Have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

* Past or current use of myopia control treatment or involvement in previous myopia control study
* Any current or seasonal use of ocular medication (eg. for allergy or chronic blepharitis).
* hypersensitivity or allergic reaction to atropine, cyclopentolate, topical anesthetics or study approved rewetting drop solutions available in local markets.
* previous history or signs of a contact lens-related corneal inflammatory event (e.g., past ulcer or scar) that may contraindicate contact lens wear.
* Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, ocular hypertension, glaucoma, history of recurrent corneal erosions, aphakia, uveitis, severe keratoconjunctivitis sicca, keratoconus, keratoconus suspect, and pellucid marginal degeneration.
* Grade 3 or greater palpebral conjunctival observations or any other Grade 2 or greater slit-lamp findings (eg. edema, corneal neovascularization, corneal staining, conjunctival injection) on the ISO 11980 classification scale.
* Any central corneal scar or corneal distortion resulting from ocular diseases or previous hard or rigid permeable contact lens wear.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in spherical equivalent | 12 months
  Change in spherical equivalent at 12 months

SECONDARY OUTCOMES:
Change in axial length | 12 months
  Change in axial length at 12 months

IPD SHARING:
Plan to Share IPD: Undecided